CLINICAL TRIAL: NCT00349713
Title: Double Blind Randomized, Controlled Phase 1 Dose Escalation Trial to Evaluate the Safety and Immunogenicity of the WRAIR AMA1 Malaria Antigen (FMP2.1) Adjuvanted in GSK's AS02A Versus Rabies Vaccine in Malaria-experienced Adults in Bandiagara, Mali
Brief Title: FMP2.1/AS02A: Rabies Vaccine Malaria-Experienced Adults in Bandiagara, Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); GlaxoSmithKline (Industry); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-031; N01AI085346-006 (NIH); N01AI085346-005 (NIH); N01AI085346-000 (NIH); 102231 ( Malaria-037) (Other: GSK); HSRRB A-12855 (Other: USAMRMC)
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-04

CONDITIONS: Malaria; Plasmodium Falciparum Malaria
Keywords: Plasmodium falciparum Malaria, Mali, adjuvant
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: 25ug FMP2.1 / AS02A (Experimental): 20 subject to receive 25ug of FMP2.1 vaccine in 0.25mL of GSK Biologicals' adjuvant AS02A
  Interventions: Biological: FMP2.1/AS02A
- Cohort 2: 50ug FMP2.1 / AS02A (Experimental): 20 subjects to receive 50ug of FMP2.1 vaccine in 0.5mL of GSK Biologicals' adjuvant AS02A
  Interventions: Biological: FMP2.1/AS02A
- Cohorts 1 and 2: Rabies vaccine (RabAvert) (Active Comparator): 20 subjects to receive Rabies vaccine (RabAvert). 10 subjects from Cohort 1 and 10 subjects from Cohort 2
  Rabies vaccine (RabAvert): RabAvert Rabies vaccine
  Interventions: Biological: FMP2.1/AS02A; Biological: Rabies vaccine (RabAvert)

INTERVENTIONS:
Biological: FMP2.1/AS02A — FMP2.1 in GSK Biologicals' AS02A
Biological: Rabies vaccine (RabAvert) — RabAvert Rabies vaccine
  Arms: Cohorts 1 and 2: Rabies vaccine (RabAvert)

SUMMARY:
Malaria is a disease that affects many people in Africa and in Mali. It is caused by germs that are spread by mosquito bites. This study will look at the safety, effectiveness, and best dose of an experimental malaria vaccine in people who are regularly exposed to malaria. Study participants will be 60 adults, 18-55 years old, who live in Bandiagara, Mali. Volunteers will get either 3 full doses of the experimental malaria vaccine, 3 half doses of the malaria vaccine, or a rabies vaccine that has been approved in Mali. (Rabies is an infection of the brain that usually causes death, and can be caught from being bitten by infected dogs or bats.) The 3 vaccinations will be given by injection into the upper arm 30 days apart. Volunteers will be enrolled in the study for approximately 12 months after the first vaccination. Volunteers will have 14 blood samples collected during the study for testing to make sure that the vaccine is not harmful and to measure the effect of the vaccine.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and reactogenicity of two dose levels of WRAIR's AMA1 malaria antigen (FMP2.1) adjuvanted in GlaxoSmithKline Biologicals' AS02A compared to rabies vaccine in malaria-experienced Malian adults aged 18-55 years inclusive. Secondary objectives are to: (1) measure the magnitude and duration of antibody response to FMP2.1; (2) measure cellular immune responses to FMP2.1 at baseline and after immunization; (3) measure the inhibition of parasite growth by the in vitro GIA; and (4) determine the specificity of the antibodies to diverse AMA1 genotypes in addition to 3D7, by measuring by ELISA, and GIA on parasites with typed AMA1. A double-blind controlled dose escalation trial will allow assessment of vaccine safety in each of three groups, one group each to receive medium and full dose levels of the experimental vaccine, and one group to receive the comparator vaccine. Thirty adults will be randomized to receive the medium dose level of FMP2.1 (n=20) or rabies vaccine (n=10) and thirty to receive the full dose level of FMP2.1 (n=20) or rabies vaccine (n=10). The division of the rabies group into two groups of ten is done to maintain blinding at each immunization time point, and all participants who receive the rabies vaccine will be analyzed as a single group. The sample size of the groups, however, will not allow detection of anything other than very large differences in the occurrence of adverse events among the three groups. The advantage of double blinding is to remove the potential for investigator and participant prejudgment about the effects of the vaccines in the reporting of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. A male or non-pregnant female aged 18-55 years inclusive at the time of screening
2. For women, willingness not to become pregnant until 1 month after the last immunization (pre-menopausal female participants will be referred to the local family planning clinic in Bandiagara, which offers several means of contraception that are approved and recommended by the Malian Ministry of Health)
3. Separate written informed consent obtained from the participant before screening and study start, respectively
4. Available and willing to participate in follow-up for the duration of study (12 months)

Exclusion Criteria:

1. Previous vaccination with any investigational vaccine or with any rabies vaccine
2. Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first study immunization, or planned use up to 30 days after the third immunization
3. Chronic administration (defined as more than 14 days) of immuno-suppressants or other immune-modifying drugs within six months prior to the first immunization. This will include any dose level of oral steroids or inhaled steroids, but not topical steroids
4. Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before the first study immunization with the exception of tetanus toxoid
5. Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
6. Any confirmed or suspected autoimmune disease
7. History of allergic reactions or anaphylaxis to immunizations or to any vaccine component
8. History of serious allergic reactions to any substance, requiring hospitalization or emergent medical care
9. History of allergy to tetracycline, doxycycline, nickel, Imidazole, chicken eggs, processed bovine gelatin, chicken protein, neomycin, or amphotericin B
10. History of splenectomy
11. Serum ALT >/=43 IU/L
12. Serum creatinine level >113 µmol /L for males and 70 µmol /L for females
13. Hgb <11 g/dL for males and <10 g/dL for females
14. WBC <4.0 x 1000/cubic mm or >13 x 1000/cubic mm
15. Absolute lymphocyte count </=1.4 x 1000 /µl
16. Thrombocytopenia < 108,000/µl
17. More than trace protein, more than trace hemoglobin or positive glucose in urine
18. Administration of immunoglobulins and/or any blood products within the three months preceding the first study immunization or planned administration during the study period
19. Suspected or known current alcohol or illicit drug abuse
20. Pregnancy or positive urine beta-HCG on the day of or prior to immunization
21. Breastfeeding
22. Simultaneous participation in any other interventional clinical trial
23. Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurological condition, or any other findings that in the opinion of the Principal Investigator (PI) may increase the risk of participating in the study
24. Other condition that in the opinion of the PI would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2004-11; Primary Completion 2005-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahamadou A. Thera, M.D., Principal Investigator — University of Bamako; Chris V. Plowe, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Bamako, Malaria Research and Training Center, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data with
  National Institute of Allergy and Infectious Diseases (NIAID)
  Walter Reed Army Institute of Research (WRAIR)
  GlaxoSmithKline
  University of Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 175 participants were screened; 115 were excluded; 60 subjects were randomized in a 2:1 ratio into 2 cohorts
Groups:
- Cohort 1: FMP2.1 / AS02A: 20 subject to receive 25ug of FMP2.1 vaccine in 0.25mL of GSK Biologicals' adjuvant AS02A
  FMP2.1/AS02A: FMP2.1 in GSK Biologicals' AS02A
- Cohort 2: FMP2.1 / AS02A: 20 subjects to receive 50ug of FMP2.1 vaccine in 0.5mL of GSK Biologicals' adjuvant AS02A
  FMP2.1/AS02A: FMP2.1 in GSK Biologicals' AS02A
Period: Overall Study
Arm/Group | Cohort 1: FMP2.1 / AS02A | Cohort 2: FMP2.1 / AS02A | Cohorts 1 and 2: Rabies Vaccine (RabAvert)
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 25ug FMP2.1 / AS02A | Cohort 2: 50ug FMP2.1 / AS02A | Cohorts 1 and 2: Rabies Vaccine (RabAvert) | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 16 | 16 | 17 | 49
Region of Enrollment [Count of Participants; unit: Participants]
  Mali | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Safety and Reactogenicity (SAEs and AEs)
Description: The primary objective was to evaluate the safety and reactogenicity of 2 dose levels of WRAIR's AMA1 malaria antigen (FMP2.1) adjuvanted in GlaxoSmithKline Biologicals' (GSK) AS02A compared to rabies vaccine in malaria-experienced Malian adults aged 18-55 years inclusive. Solicated AEs were recorded for the 7 day surveillance period after each vaccination. Unsolicited AEs were recorded for 30 days after each vaccination.
Time Frame: 12 months
Population: Summary of Adverse Events by Group and Immunization Group
Measure: Number; unit: Number of events
Arm/Group | Cohort 1: 25ug FMP2.1 / AS02A | Cohort 2: 50ug FMP2.1 / AS02A | Cohorts 1 and 2: Rabies Vaccine (RabAvert)
Number analyzed (Participants) | 20 | 20 | 20
Number of events
  Solicited: Injection Site Pain | 45 | 53 | 22
  Solicited: Injection Site Swelling | 37 | 35 | 11
  Solicited: Arm Motion Limitation | 5 | 3 | 0
  Solicited: Elevated Temperature | 6 | 6 | 1
  Solicited: Headache | 7 | 17 | 9
  Solicited: Chills | 4 | 2 | 4
  Solicited: Malaise | 4 | 5 | 3
  Solicited: Nausea | 4 | 1 | 1
  Solicited: Arthralgia | 0 | 2 | 1
  Solicited: Myalgia | 3 | 6 | 3
  Solicited: Erythema | 0 | 0 | 0
  Unsolicited: Cold | 21 | 10 | 7
  Unsolicited: Headaches | 11 | 11 | 5
  Unsolicited: Coughing | 8 | 3 | 3
  Unsolicited: Flu | 6 | 3 | 3
  Unsolicited: Wound | 3 | 2 | 4
  Unsolicited: Myalgia | 2 | 2 | 4
  Unsolicited: Scratch | 1 | 2 | 3
  Unsolicited: Diarrhea | 1 | 2 | 3
  Unsolicited: Pruritus | 1 | 4 | 1

2. Secondary Outcome: Antibody Response to FMP2.1 Over Time
Description: Measurement of anti-AMA1 antibody titers over time
Time Frame: 90 Days
Population: Anti-AMA1 Antibody titers on days, 0, 14, 30, 44, 60, 74, and 90
Measure: Mean (Standard Deviation); unit: Antibody Titers
Arm/Group | Cohort 1: 25ug FMP2.1 / AS02A | Cohort 2: 50ug FMP2.1 / AS02A | Cohorts 1 and 2: Rabies Vaccine (RabAvert)
Number analyzed (Participants) | 20 | 20 | 20
Antibody Titers
  Day 0 | 53295.3 (76881) | 56779.4 (53811.2) | 59852 (101952.4)
  Day 14 | 62963.8 (77633.3) | 120677.4 (104675.9) | 63697.6 (119009.9)
  Day 30 | 68251.2 (87406.5) | 101464.5 (99045.2) | 51436.1 (95888.9)
  Day 44 | 101478.2 (139781.1) | 159449.2 (152111.2) | 62498.3 (115667.3)
  Day 60 | 103966.8 (117998.7) | 187453.9 (162090.9) | 77418.1 (147844.9)
  Day 74 | 128323.7 (109759) | 227692.0 (236420.5) | 82794.3 (173534.6)
  Day 90 | 87684.2 (99596.7) | 162739.7 (182897.2) | 52575.5 (99568.0)

3. Secondary Outcome: Anti-AMA1 Log Antibody Titers Over Time
Description: Summary of Anti-AMA1 Log Antibody titers on days 0, 14, 30, 44, 60, 74 and 90
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: log antibody titers
Arm/Group | Cohort 1: 25ug FMP2.1 / AS02A | Cohort 2: 50ug FMP2.1 / AS02A | Cohorts 1 and 2: Rabies Vaccine (RabAvert)
Number analyzed (Participants) | 20 | 20 | 20
log antibody titers
  Day 0 | 4.3 (0.7) | 44.4 (0.9) | 4.2 (0.8)
  Day 14 | 4.5 (0.6) | 4.8 (0.6) | 4.1 (0.8)
  Day 30 | 4.5 (0.6) | 4.7 (0.6) | 4.1 (0.8)
  Day 44 | 4.7 (0.5) | 5.0 (0.5) | 4.1 (0.8)
  Day 60 | 4.8 (0.5) | 5.1 (0.5) | 4.2 (0.8)
  Day 74 | 4.9 (0.4) | 5.2 (0.4) | 4.1 (0.8)
  Day 90 | 4.8 (0.4) | 5.0 (0.4) | 4.0 (0.9)

4. Secondary Outcome: Geometric Mean Antibody Titers Over Time
Description: Measurement of geometric mean antibody titers on days 0, 14, 30, 44, 60, 74 and 90
Time Frame: 90 Days
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean of Antibody Titers
Arm/Group | Cohort 1: 25ug FMP2.1 / AS02A | Cohort 2: 50ug FMP2.1 / AS02A | Cohorts 1 and 2: Rabies Vaccine (RabAvert)
Number analyzed (Participants) | 20 | 20 | 20
Geometric Mean of Antibody Titers
  Day 0 | 19161.2 [8569.5 to 42843.9] | 23499.7 [9078.9 to 60825.6] | 14354.8 [5859.8 to 35164.9]
  Day 14 | 30795.3 [16398.1 to 57829.4] | 69751.6 [37929.2 to 128272.7] | 13856.7 [5568.2 to 34483.1]
  Day 30 | 31804.9 [16571.8 to 61040.8] | 55085.8 [29386.5 to 103260.1] | 12690.7 [5296.6 to 30407.1]
  Day 44 | 55246.5 [33102.4 to 92204.0] | 100589.6 [61275.4 to 165127.7] | 13941.2 [5719.8 to 33979.9]
  Day 60 | 61438.6 [36763.7 to 102674.5] | 119191.3 [71967.1 to 197403.6] | 16030.5 [6502.6 to 39518.8]
  Day 74 | 89856.7 [57817.9 to 139649.3] | 150738.4 [97729.2 to 232500.5] | 14064.5 [5534.1 to 35743.6]
  Day 90 | 60967.1 [41140.3 to 90348.9] | 102813.0 [65715.6 to 160852.4] | 10425.1 [4079.6 to 26640.2]

5. Secondary Outcome: Subjects With 2- and 4-fold Increases in Anti-FMP2.1 Antibody Levels Over Time
Description: Proportion of Subjects with 2- and 4-fold increases in Anti-FMP2.1 Antibody levels on days 14, 30, 44, 60, 74 and 90
Time Frame: 90 Days
Measure: Number; unit: number of participants with increase
Arm/Group | Cohort 1: 25ug FMP2.1 / AS02A | Cohort 2: 50ug FMP2.1 / AS02A | Cohorts 1 and 2: Rabies Vaccine (RabAvert)
Number analyzed (Participants) | 20 | 20 | 20
number of participants with increase
  Day 14 2-fold increase | 5 | 9 | 0
  Day 14 4-fold increase | 1 | 5 | 0
  Day 30 2-fold increase | 2 | 4 | 0
  Day 30 4-fold increase | 2 | 4 | 0
  Day 44 2-fold increase | 3 | 6 | 0
  Day 44 4-fold increase | 3 | 6 | 0
  Day 60 2-fold increase | 6 | 7 | 0
  Day 60 4-fold increase | 6 | 7 | 0
  Day 74 2-fold increase | 9 | 11 | 0
  Day 74 4-fold increase | 9 | 11 | 0
  Day 90 2-fold increase | 6 | 7 | 0
  Day 90 4-fold increase | 6 | 7 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Cohort 1: 25 ug FMP2.1 / AS02: 25 ug FMPs.1 / AS02
- Cohort 2: 50 ug FMP2.1 / AS02A: 50 ug FMP2.1 / AS02A
- Cohort 3: Rabies Vaccine (RabAvert): Rabies vaccine, All events reports instead of AE's per vaccination group 20 subjects (10 from Cohort 1 and 10 from Cohort 2)
Arm/Group | Cohort 1: 25 ug FMP2.1 / AS02 | Cohort 2: 50 ug FMP2.1 / AS02A | Cohort 3: Rabies Vaccine (RabAvert)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 20/20 | 20/20 | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 25 ug FMP2.1 / AS02 (N=20) | Cohort 2: 50 ug FMP2.1 / AS02A (N=20) | Cohort 3: Rabies Vaccine (RabAvert) (N=20)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Abrasion from scratching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute injection site pain (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0)
Acute lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute left inferior deltoid pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute viral rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic cold symptoms (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic conjunctivitis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anorxia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Bacterial conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bilateral ocular pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bilateral pruritus of forearms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bilious vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blood streak in stool (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Boil (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bullous pruritic lesions of upper extremities (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Burning muscular pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Burning with urination (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Chills (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 1 (1)
Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (7)
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 5 (5) | 0 (0)
Cold symptoms with productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Coxalgy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dental abscess tooth #21 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dental cavity tooth #18 (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Dermatomycosis of inguinal folds (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Diffuse headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1) | 0 (0)
Dysentery (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Edema of left anterior forearm (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated blood pressure = 150/90 mmHg (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated temperature (Investigations) | 0 (0) | 0 (0) | 2 (2)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Epistaxis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Erythema extending from injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Evening headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Excessive sweating (General disorders) | 0 (0) | 1 (1) | 0 (0)
Extrasystol (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Eye tearing and itching (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Facial sweating (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile at 37.5 C (General disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile to 37.8 C (General disorders) | 0 (0) | 1 (1) | 0 (0)
Heart racing (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 6 (6) | 4 (4) | 0 (0)
Flu (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Flu like symptoms (General disorders) | 11 (11) | 8 (8) | 0 (0)
Foreign body in eye causing tearing (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Frontal headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Frontal sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Generalized pruritus and skin papules (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Groin elongation (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Gum pain following tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 20 (20) | 17 (17) | 5 (5)
Headache in frontal region (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache in temporal region (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Headaches (Nervous system disorders) | 3 (3) | 7 (7) | 5 (5)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hives (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypochondrium pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Induced injection site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injection site edema (grade 1) (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 0 (0)
Injection site edema (grade 2 (Injury, poisoning and procedural complications) | 20 (20) | 9 (9) | 0 (0)
Injection site edema (grade 3) (Injury, poisoning and procedural complications) | 9 (9) | 20 (20) | 0 (0)
Injection site pain (grade 1) (Injury, poisoning and procedural complications) | 20 (20) | 20 (20) | 1 (1)
Injection site pain (grade 2) (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
Injection site pain with pulsatile sensation (grade 1) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injection site pain extending to left elbow (grade 1) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injection site pain extending to left shoulder (grade 1) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injection site pain with movement (grade 1) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injection site pulsation (grade 1) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 8 (8)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Isolated pruritus of the umbilical region (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis left eye (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Left food punture wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Left foot scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Left foot wound on lateral, external aspect (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Left otalgia (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Left pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Left rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Left upper premolar tooth pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Limitation of arm movement (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 0 (0)
Liquid diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Lombalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Loss of balance with movement (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lower back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Malaise (General disorders) | 6 (6) | 7 (7) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mucsle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle pain of abdominal muscles and at venipuncture site (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular pain of right lower extremity following trauma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 11 (11) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0)
Needle stick injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Nighttime cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nighttime wet cough triggered by cigarette smoke (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Non-pruritic papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular affection (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Oropharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pain at venipuncture site (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Pain in right hypochondium (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in anterior left forearm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain of right knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain of right hypochondrium (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain with shaking of the right hypochondrium (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain with urination (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Painful dental cavity (tooth extraction) (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Palpitation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Papule of the posterior ankle and inferior left abdominal flank (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Papule on mid-flank of right abdomen (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Papule pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Papule unpruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Papules + pruritus following an insect bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal vertigo (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Physical weakness (General disorders) | 2 (2) | 3 (3) | 0 (0)
Pityriasis versicolor (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Positive urine pregnancy test (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
post-operative pain at wound site (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic edema of forehead (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic pain of the right elbow and wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic right foot pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Premature/ectopic heart beat (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Presence of blood in stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pruritic papules (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritis of internal face of thighs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritis papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritis with papules and excoriation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritis with skin abrasions from scratching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pulled groin muscle (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Purulent conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 9 (9) | 0 (0)
Rhinitis of mucous membranes (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinobronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Rhinopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Rhinosinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Right ankle pain after dislocation since 2002 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Right ankle traumatic wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Right eye conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Right eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Right eye pterygium (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Right index finger traumatic wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Right inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Right leg traumatic wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Right lumbar pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Right otitis (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Right tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Right wrist scratch on posterior aspect (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ringing in the ears (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Scratch of anterior/external aspect of the thigh (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sensation of arm heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sensation of head heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Sense of pulsation at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sinisitis + Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subjective evening fever (General disorders) | 2 (2) | 2 (2) | 0 (0)
Super infected wounds on left leg (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Surgical hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Sweats (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling of right thumb (General disorders) | 0 (0) | 1 (1) | 0 (0)
Syndrome of tissue hyperfusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Syndrome typhic (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Tachycardia at 100beats/min (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Temperature = 37.5C (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thumb inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Torticollis (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Transient loss of balance (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Traumatic leg wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic pain of left toes (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic wound of right ring fingure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic wound of the middle finger (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic wound of the right knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Typhoid syndrome (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Uncomplicated malaria episode (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urethral discharge (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 5 (5)
Vertigo (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Viral rhinopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Visual floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vulvitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Whitish leukorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No